CLINICAL TRIAL: NCT04564573
Title: The Impact of Systemic Antidepressant Treatments in Early Stage on Neurocognitive Function of Euthymic Patients With Bipolar Depression
Brief Title: Antidepressant Treatments and Cognitive Function of Bipolar Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJAH2020-18
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-09

CONDITIONS: Bipolar Disorder; Cognition
Keywords: antidepressant treatment; euthymic state; neurocognitive function; bipolar depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Ten milliliters of venous blood are adopted from each participant into a free-anticoagulant vacuum tube. The blood will be immediately centrifuged at 4,000 g for 10 min, and serum is kept frozen at -80 ºC until analysis. NSE levels are measured with electrochemiluminescence assay, using a commercial kit conforming to the manufacturer instructions and data will be shown in ng/ml.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antidepressant treatment group: participants who had received systemic antidepressant (consecutive treatment with adequate antidepressants for 6 weeks at least)treatment in the early stage (from initial depressive onset to first manic/hypomani episode).
- non-antidepressant treatment group: participants who had not received systemic antidepressant (consecutive treatment with adequate antidepressants for 6 weeks at least)treatment in the early stage (from initial depressive onset to first manic/hypomani episode).

SUMMARY:
Patients with bipolar disorder (BD) have a wide range of neurocognitive dysfunction, which lead to impaired psychosocial function and reduced quality of life. Therefore, improving neurocognitive function has become an important goal of BD treatment. Aiming at this, some clinical studies have been performed but failed to illustrate significant positive efficacies of pharmacological therapy or non-pharmacological therapy, which could attribute in part to insufficient understanding on the risk factors that affect the neurocognitive function of BD patients. Delayed diagnosis of BD is so common that a lot of patients receive long-term antidepressant treatment before of diagnosis of unipolar depression. There is controversy about whether antidepressant treatment in early stage would affect the neurocognitive function of BD patients. In view of the high prevalence of delayed diagnosis and the use of antidepressants, it is of great scientific significance and clinical value to clarify this matter and other factors that may potentially affect the neurocognitive function of BD patients.

DETAILED DESCRIPTION:
Subjects will not be engaged with any interventions in this study. Two senior psychiatrists are in attendance of screening the patients with the inclusion/exclusion criteria, and then all patients who meet both criteria and are willing to participate in this study will sign the informed consent before enrollment. The participants will be divided into AT or NT group according to their history of antidepressant treatment in early stage, which is done by the two senior psychiatrists. Then these senior psychiatrists will also collect additional study parameters, such as age, sex, nation, age of onset, and score of Premorbid Adjustment Scale (PAS). Furthermore, the information about history of treatments and diagnosis will be further confirmed with medical documentary and patients' guardians. Afterwards, other investigators will finish the rating work of the rest of scales. The whole procedure should be done within 180 min. Finally, ten milliliters of venous blood are adopted for measuring NSE

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of BD diagnosed according to the Diagnostic and Statistical Manual of Mental disorders, Fourth Edition (DSM-IV-TR) diagnosed with Structured Clinical Interview for DSM-IV (SCID); a current state of euthymia is defined by both scores of Montgomery-Åsberg Depression Scale (MADRS) and Young Manic Rating Scale (YMRS) <7, lasting for 4 weeks at least before recruitment
2. Initiated with a depressive episode
3. Aged between 18~50 years
4. Patients comply with all procedures of study
5. Participants must sign the informed consent

Exclusion Criteria:

1. A history of psychiatric symptoms
2. A comorbidity of attention deficit and hyperactivity disorder (ADHD)
3. Neurological trauma or neurological diseases which could cause cognition injury
4. History of substance dependence/abuse
5. Received modified electroconvulsive therapy (MECT) in the past 12 months
6. Severe physical disease affecting cognitive function or increasing peripheral NSE
7. Recent drug use that affects cognition, such as tricyclic antidepressants, anticholinergic drugs, amphetamines, etc.
8. IQ <70
9. Use benzodiazepines 4 hours before scale evaluation

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: This study will consist of a sample of 124 patients with bipolar disorder who initiated with a depressive episode and being a euthymic state for 4 weeks at least before enrollment.All participants are divided into two groups according to whether they had received systemic antidepressant treatment or not in the early stage.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Subjective cognitive measures | before 11AM
  cognitive complaints in Bipolar Disorder Rating Assessment (COBRA)
Objective cognitive measures | before 11AM
  the Stroop Color and Word Test (SCWT), the categorical verbal fluency test (CVFT) (animal naming), and the Trail Making Test Part B (TMT-B), the Digital Span Forward and Backward subtest (DSFB) and the Digit Symbol Coding subtest (DSC) of the Wechsler Adult Intelligence Scale-Revised by China (WAIS-RC) and Trail Making Test Part A (TMT-A), the Visual Reproduction subtest (VRP) and the Visual Recognition subtest (VRC) of the Wechsler Memory Scale-Revised (WMS-R)

SECONDARY OUTCOMES:
Global Assessment Function (GAF) | before 11AM
  to assess patients' functions psychologically, socially and professionally
Methods Checklist on Quality of Life issued by World Health Organization-Brief version,WHOQOL-BRIEF | before 11AM
  to assess the quality of life
Peripheral neuron-specific enolase (NSE) | before 11.30AM
  to test the potential injury of neuron

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index,PSQI | before 11AM
  to evaluate the quality of sleep
Positive and Negative Affect Scale,PANAS | before 11AM
  to detect the change in positive and negative affect

CONTACTS AND LOCATIONS:
Overall Officials: Chenghao Yang, Doctor, Principal Investigator — Tianjin Anding Hospital
Locations (1):
- Tianjin Anding Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes
Request based on researcher's consent
Supporting Information: Study Protocol, SAP, ICF
Time Frame: the data will be available openly after the study finished with no termination.

REFERENCES:
- [Derived] Yang H, Liu Y, Yang C, Lin X. The effect of systemic antidepressant treatments in early stage on neurocognitive function of euthymic bipolar patients initiated with a depressive onset: An observational, cross-sectional, single-blind study protocol. Brain Behav. 2021 Oct;11(10):e2360. doi: 10.1002/brb3.2360. Epub 2021 Sep 14. PMID 34520638